CLINICAL TRIAL: NCT06310850
Title: The Effect of Preprocedural Subanesthetic Ketamine for Pain and Anxiety in Patients During Thoracic Epidural Catheterization: A Randomized Trial
Brief Title: The Effect of Preprocedural Subanesthetic Ketamine on Pain and Anxiety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Onur Kucuk, Principal Investigator, Ankara Ataturk Sanatorium Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KEAH-238
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Epidural Catheterization; Thoracic; Procedural Pain
Keywords: ketamine; pain; anxiety; subanesthetic
MeSH Terms: conditions — Pain, Procedural; Pain; Anxiety Disorders | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized, prospective study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Placebo (Placebo Comparator): intravenous placebo
  Interventions: Other: Placebo
- Group Ketamine (Active Comparator): intravenous ketamine 0.15 mg kg-1
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Patients will be administered 0.15 mg kg-1 intravenous ketamine (The sample provided contains equal proportions of two enantiomers, S and R ketamine hydrochloride.) 3 minutes before thoracic epidural catheter placement.
  Arms: Group Ketamine
Other: Placebo — Intravenous saline will be administered to patients 3 minutes before the thoracic epidural catheter is placed.
  Arms: Group Placebo

SUMMARY:
The thoracic epidural catheterization (TEC) can be both uncomfortable and fearful for patients when done awake with the thought that the procedure may be painful. The aim of this study was to assess the effect of subanesthetic intravenous ketamine administration on pain and anxiety during the TEC procedure.

DETAILED DESCRIPTION:
The study aimed to assess the impact of subanesthetic intravenous ketamine administration on pain and anxiety during Thoracic Epidural Catheterisation (TEC) procedure, which can be uncomfortable and frightening for patients when performed awake due to the possibility of pain.

After receiving approval from the clinical research ethics committee of Keçiören Education and Research Hospital (KEAH; ID:238), this prospective and randomized study will include 60 adult patients with ASA physical status I-III who are scheduled for elective thoracic surgery via thoracotomy. The study will randomly assign patients into two groups: Group P (n=30) receiving an intravenous placebo and Group K (n=30) receiving intravenous (IV) 0.15 mg kg-1 ketamine. Randomisation will be performed using a computerised table of random numbers.

Patients with chronic pain, bleeding disorders, drug use, liver disease, severe metabolic and endocrine problems, a history of ketamine or local anaesthetic allergy, infection at the site of intervention, or refusal of TEC will be excluded. Patients who report acute pain during preoperative evaluation, have a TEC time of more than five minutes (from needle insertion to catheter insertion), and require more than two Tuohy needle attempts will be excluded. Vital parameters and anxiety levels of each patient will be recorded before premedication. Anxiety (VAS-A) and pain (VAS-P) scores will be measured using the visual analogue scale. Patients will be transported to the operating theatre 20 minutes after premedication. Intravenous administration of 0.15 mg/kg IV ketamine or placebo will take place 3 minutes before TEC placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective thoracic surgery via thoracotomy
* Patients with ASA physical status I-III

Exclusion Criteria:

* Describing chronic pain,
* Have a bleeding disorder,
* Having a history of analgesia drug use,
* Have a history of liver disease,
* Have serious metabolic and endocrine problems,
* Have a history of allergy to ketamine and local anesthetics,
* Have an infection in the intervention area,
* Rejecting thoracic epidural catheter,
* Describing acute pain in any part of the body during the preoperative evaluation,
* Thoracic epidural catheter duration greater than five minutes (time from needle entry to catheter placement)
* Patients requiring more than two Tuohy injection attempts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 1 day (5 times)
  For anxiety, on a 100 mm scale, 0 mm was defined as no anxiety, whereas 100 mm was as unbearable anxiety (VAS-A). A similar scoring method was used to assess pain intensity. 0 mm was defined as no pain and 100 mm as unbearable pain (VAS-P).

CONTACTS AND LOCATIONS:
Overall Officials: Onur KÜÇÜK, specialist, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No